CLINICAL TRIAL: NCT05834972
Title: Ultrasound-guided Versus Landmark-guided Percutaneous Dilational Tracheostomy in Pediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, Cengiz Kılıçarslan, Medical Doctor, Aksaray University
Other Study IDs: 34-SBKAEK-2023-05-05
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Tracheostomy Complication; Tracheostomy Hemorrhage; Airway Trauma; Percutaneous Tracheostomy
Keywords: percutaneous dilatational tracheostomy; ultrasound guided tracheostomy; landmark guided tracheostomy; pediatric patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Landmark-guided percutaneous dilatational tracheostomy: All patients will be enrolled two times. First, an experienced anesthesiologist will examine the neck anatomy and mark the second or third tracheal ring using the traditional landmark-guided technique, and the duration will be recorded. Then, the same anesthesiologist will examine the neck anatomy and mark the second or third tracheal ring using the ultrasound (USG)-guided approach, and the duration will be recorded. The distance between these two aforementioned markings will be measured and recorded. The first marking determined by the landmark method will be looked at with USG and where it corresponds anatomically will be recorded. Also, the vascular and glandular structures of the area and potential complications will be noted.
- Ultrasound-guided percutaneous dilatational tracheostomy: All patients will be enrolled two times. First, an experienced anesthesiologist will examine the neck anatomy and mark the second or third tracheal ring using the traditional landmark-guided technique, and the duration will be recorded. Then, the same anesthesiologist will examine the neck anatomy and mark the second or third tracheal ring using the ultrasound (USG)-guided approach, and the duration will be recorded. The distance between these two aforementioned markings will be measured and recorded. The first marking determined by the landmark method will be looked at with USG and where it corresponds anatomically will be recorded. Also, the vascular and glandular structures of the area and potential complications will be noted.
  Interventions: Device: Ultrasound-guided percutaneous dilatational tracheosyomy

INTERVENTIONS:
Device: Ultrasound-guided percutaneous dilatational tracheosyomy — All of the participants will be examined two times. First, the landmark-guided technique will be performed. Then, the ultrasound-guided technique will be performed.
  Other Names: Landmark-guided percutaneous dilatational tracheosyomy
  Groups: Ultrasound-guided percutaneous dilatational tracheostomy

SUMMARY:
Percutaneous dilatational tracheostomy is one of the most common procedures performed in pediatric intensive care units. The investigators aimed to compare traditional landmark-guided percutaneous dilatational tracheostomy (PDT) and ultrasound-guided percutaneous dilatational tracheostomy in pediatric patients in terms of location, duration, and potential complications related to the procedure.

DETAILED DESCRIPTION:
Tracheostomy, one of the most common procedures performed in intensive care units (ICU), refers to creating a stoma in the anterior wall of the trachea to maintain airway security. Tracheostomy can be formed via a surgical or percutaneous dilatational technique (1). The surgical technique requires the transportation of the patient to the operating theatre, while the percutaneous dilatational technique can be performed in the ICU. Thus, ICU practitioners commonly prefer the percutaneous dilatational technique.

Percutaneous dilatational tracheostomy can be performed via three approaches: landmark, ultrasound (USG), or bronchoscopy guided. Although landmark-guided PTD is a practical approach, there are growing concerns regarding the location of the second and third tracheal rings and injuries to vascular structures and the thyroid gland. USG may be helpful to establish the anatomy of the airway and the vascular and glandular structure of the area.

The investigators aimed to compare traditional landmark-guided percutaneous dilatational tracheostomy and USG-guided percutaneous dilatational tracheostomy in pediatric patients in terms of location, duration, and potential complications related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* healthy pediatric patients
* between 5 and 13 years old

Exclusion Criteria:

* neck anomalies
* syndromic patients

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy pediatric patients between 5 and 13 years old and admitted to the operating theatre and sedated will be included after the consent of their parents or legal guardians.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-25 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
Anatomical accuracy of the entry site for percutaneous dilatational tracheostomy | 20 minutes
  Identification of the second and third tracheal ring

SECONDARY OUTCOMES:
Detection of potential complications of the airway entry point determined by the traditional method | 20 minutes
  Proximity of the airway entry point determined by the traditional method to vascular and glandular structures
The time taken by the landmark-guided and ultrasound-guided techniques | 20 minutes
  Time taken to determine the airway entry point with landmark-guided and ultrasound-guided techniques

CONTACTS AND LOCATIONS:
Overall Officials: Cengizhan Kilicaslan, MD, Principal Investigator — Pediatrician
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
We will share the protocol, measurement tools that we will use, and the statistical analysis plan of the study.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available after publication.
Access Criteria: The data will be uploaded to clinicialtrials.gov

REFERENCES:
- [Background] Gobatto ALN, Besen BAMP, Cestari M, Pelosi P, Malbouisson LMS. Ultrasound-Guided Percutaneous Dilational Tracheostomy: A Systematic Review of Randomized Controlled Trials and Meta-Analysis. J Intensive Care Med. 2020 May;35(5):445-452. doi: 10.1177/0885066618755334. Epub 2018 Feb 7. PMID 29409380